CLINICAL TRIAL: NCT06450249
Title: Effects of the Humanitude® Care Methodology on Improving Health Professionals' Perception of Competence and Emotional State
Brief Title: Effects of the Humanitude® Care Methodology on Health Professionals' Perception
Acronym: Humanitude
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RNIPH-2021-23
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Delivery of Health Care; Education, Medical; Caregiver
Keywords: Humanitude; Care methodology; Agitated behavior; Quality of care; Health professional; Well being; Medical education
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals: Healthcare professionals working in Continuous Care Units before and after participation in Humanitude® Care Methodology (HCM) training sessions in the Ile-de-France region in France
  Interventions: Behavioral: Humanitude® Care Methodology (HCM) training sessions; Behavioral: Self-administered questionnaire

INTERVENTIONS:
Behavioral: Humanitude® Care Methodology (HCM) training sessions — During a five-day training session healthcare professionals are trained to the HCM within their own care unit
Behavioral: Self-administered questionnaire — The self-administered questionnaire will be completed before and after participation in Humanitude® Care Methodology training sessions

SUMMARY:
Healthcare professionals providing care for institutionalized older patients must deal with agitated behavior daily. Such behavior alters the patient's quality of life and generates stress for the caregiver. Humanitude® Care Methodology is an alternative to pharmaceutical approaches that has demonstrated benefits on care delivery. The present study aims to investigate the effects of this method on healthcare professionals' perception of competence and emotional state when dealing with difficult care situations.

DETAILED DESCRIPTION:
This is a retrospective, multicentric, before / after study. Data collected from a self-administered questionnaire to caregivers working in 32 Continuous Care Units before and after participation in Humanitude® Care Methodology training sessions in the Ile-de-France region in France will be analyzed. Data on the participants' perception of their own care competence and their emotional state when confronted with several difficult care situations will be collected. Participants' well-being at work and adhesion to the Humanitude® Care Methodology will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers taken part in a Humanitude® training course
* Caregivers agreeing to complete pre- and post-training questionnaires

Exclusion Criteria:

* Caregiver not completing the questionnaire at one of the 2 stages of the assessment (before or after)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Professionals trained in the principles and techniques of Humanitude®. For each training session, these professionals are invited to complete a questionnaire at the beginning and end of the course. These questionnaires are part of the training organization's quality approach and are designed to assess the impact of the training.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
4-point scale for evaluation of Caregivers' feelings | 5 days
  Caregivers are asked to comment on their feelings, on a 4-point scale (anxiety; apprehension; serenity; pleasure) when they enter in a resident's room before and after the training.

SECONDARY OUTCOMES:
4-point scale for evaluation of caregivers'competence | 5 days
  To collect caregivers' feelings of competence, they are asked to give their opinion on how capable they felt of looking after a resident, on a 4-point scale (not at all capable; not very capable; capable; very capable) when they entered the room of a resident
3-point scale for evaluation of caregivers' trust in their colleagues | 5 days
  The degree of trust which caregivers place in their colleagues on a daily basis is assessed on a 3-point scale : no; it's not always up to me; yes).
Scale for evaluation of caregivers' degree of pleasure in coming to work | 5 days
  The degree of pleasure in coming to work is assessed on a scale from 0 (not at all) to 10 (a lot).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Buttitta, PhD, Principal Investigator — GHICL
Locations (2):
- France (2):
  - GHICL, Lille, Nord
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille